## **RESULTS**

This study was prospectively conducted on 250 women recruited from ElShatby university maternity hospital delivery ward; they were randomized into two groups group (A) and group (B) by closed envelop randomization.

Group (A) was undergo cesarean section with bladder dissection.

Group (B) was undergo cesarean section without bladder dissection.

### I. Comparison between patients in group I and group II regarding age.

The age in group I ranged from 16-42 years with mean value  $26.12\pm6.34$  and in group II ranged from 15-41 years with mean value  $24.66\pm5.59$ . There was no statistically significant difference between the two studied groups regarding age (P= 0.067) (Table 1, Fig. 14)

Table (1): Comparison between the two studied groups regarding age.

| | Group I | Group II |
|-------------|---------|----------|
| Age (years) | | |
| Range | 16-42 | 15-41 |
| Mean | 26.12 | 24.66 |
| SD | 6.34 | 5.59 |
| T test | 1.68 | |
| P value | 0.067 | |

Group I. cesarean section with bladder dissection

Group II: cesarean section without bladder dissection

t-test = student t-test



Figure (14): Comparison between the two studied groups regarding age.

#### II-Comparison between two groups as regard obstetric history

Gravidity in group I had mean value 1.44±1.03 and in group II had mean value 1.312±0.737. Parity in group I had mean value 0.136±0.68 and in group II had mean value 0.192±0.73. It was found that most of cases had no abortion in two studied groups 97(77.6%) and 99(79.2%) respectively. No ectopic cases was higher with 125(100%) and 124(99.2%) respectively. Gestational age had mean value 37.41±2.37 and in group II had mean value 36.99±2.50.

There were no statistically significant differences between the two studied groups regarding gravidity (P = 0.133), parity (P = 0.069), abortion (P = 0.465), ectopic (P = 0.159) and gestational age (P = 0.175). (Table 2, Fig. 15)

Table (2): Comparison between the two studied groups regarding obstetric history.

| Obstetric history | Group I | Group II | T test<br>P value |
|-------------------|-------------|-------------|-------------------|
| Gravidity | | | |
| Range | 1-9 | 1-6 | 0.133 |
| Mean | 1.44 | 1.312 | 0.133 |
| SD | 1.03 | 0.77 | |
| Parity | | | |
| Range | 0-6 | 0-4 | 0.069 |
| Mean | 0.142 | 0.192 | 0.009 |
| SD | 0.68 | 0.73 | |
| Abortion | | | |
| No | 97 (77.6%) | 99 (79.2%) | 0.465 |
| 1-2 | 27 (21.6%) | 23 (18.4%) | 0.403 |
| >2 | 1 (0.8%) | 3 (2.4%) | |
| Ectopic | | | |
| No | 125(100.0%) | 124 (99.2%) | 0.159 |
| Yes | 0.0 (0.0%) | 1 (0.8%) | |
| Gestational age | | | 0.175 |

| Range | 34-41 | 33-41 |
|-------|-------|-------|
| Mean | 37.41 | 36.99 |
| SD | 2.37 | 2.50 |

Group I. cesarean section with bladder dissection t-test = student t-test Group II: cesarean section without bladder dissection p was significant if  $\leq 0.05$ 









**Figure (15):** Comparison between the two studied groups regarding obstetric history.

#### III-Comparison between two groups as regard uterine position

AVF position in both groups was higher 108(86.4%) and 116(92.8%) respectively followed by RVF position with 15(12%) and 8(6.4%) respectively, erect position was equal in both groups with 1(0.8%). There was statistical significant increase in group I than group II regarding the RVF position (P=0.03). (Table 3, Fig. 16)

Table (3): Comparison between the two studied groups regarding the uterus position.

| Uterus | Group I | | Gro | up II | P value |
|----------|---------|------|-----|-------|---------|
| position | No | % | No | % | |
| AVF | 109 | 87.2 | 116 | 92.8 | 0.265 |
| RVF | 15 | 12.0 | 8 | 6.4 | 0.03* |
| Erect | 1 | 0.8 | 1 | 0.8 | 1.0 |

Group I. cesarean section with bladder dissection

Group II: cesarean section without bladder dissection

 $X^2$  = Chi square-test

<sup>\* =</sup> Significant at level 0.05



Figure (16): Comparison between the two studied groups regarding the uterus position.

#### IV-Comparison between two groups as regard incidence of niche

Niche is defined as an anechoic space at least 2 mm depth at the presumed site of the caesarean section scar.

The incidence of niche was higher in group I, yet it did not reach statistical significance. (P=0.087). (Table 4, Fig. 17)

Table (4): Comparison between the two studied groups regarding incidence of niche

| Incidence of niche | Group I | | Group II | |
|--------------------|---------|------|----------|------|
| | No | % | No | % |
| Absent | 89 | 71.2 | 99 | 79.2 |
| Present | 35 | 28.0 | 26 | 20.8 |
| $X^2$ | 1.94 | | | |
| P value | 0.087 | | | |

Group I. cesarean section with bladder dissection

Group II: cesarean section without bladder dissection

 $\chi^2$  = Chi square-test



Figure (17): Comparison between the two studied groups regarding incidence of niche

#### V- Comparison between the two groups regarding niche characteristics

Length in group I ranged from 0.3-1.1 with mean value  $0.707\pm0.23$  and in group II ranged from 0.32-1.4 with mean value  $0.570\pm0.21$ . Width in group I ranged from 0.35-1.3 with mean value  $0.737\pm0.26$  and in group II ranged from 0.4-1.12 with mean value  $0.640\pm0.19$ . There was statistical significant increase in group I than group II regarding length and width (P=0.010, 0.046). There were no statistical significant differences between the two studied groups regarding depth, AMT and RMT (P=0.421, 0.441, 0.378). (Table 5, Fig. 18)

Table (5): Comparison between the two studied groups regarding niche characteristics.

| Niche characteristics | Group I | Group II | T test<br>P value |
|-----------------------|-----------|-----------|-------------------|
| Length (cm) | | | |
| Range | 0.3-1.1 | 0.32-1.4 | 0.010* |
| Mean | 0.707 | 0.570 | 0.010* |
| SD | 0.23 | 0.21 | |
| Width (cm) | | | |
| Range | 0.35-1.3 | 0.4-1.12 | 0.046* |
| Mean | 0.737 | 0.640 | 0.046* |
| SD | 0.26 | 0.19 | |
| Depth (cm) | | | |
| Range | 0.21-0.80 | 0.20-0.49 | 0.421 |
| Mean | 0.331 | 0.317 | 0.421 |
| SD | 0.15 | 0.09 | |
| AMT | | | |
| Range | 0.85-1.6 | 0.92-1.39 | 0.441 |
| Mean | 1.109 | 1.115 | 0.441 |
| SD | 0.16 | 0.14 | |
| RMT | | | |
| Range | 0.24-1.4 | 0.34-0.92 | 0.378 |
| Mean | 0.716 | 0.701 | 0.376 |
| SD | 0.21 | 0.15 | |

Group I. cesarean section with bladder dissection

Group II: cesarean section without bladder dissection

t-test = student t-test

\* = Significant at level 0.05







Figure (18): Comparison between the two studied groups regarding niche characteristics.

## VI- Comparison between the two groups regarding post delivery complain

The incidence of post-delivery complaint (HMB, Intermenstrual spotting and post coital bleeding) after 6 months was more in group I than group II, but it did not reach statistical significance. The most common complaint was spotting 8(61.5%) v.s 4(50%) followed by post coital bleeding 3(23.1%) v.s 2(25%).

So ,There was no statistical significant difference between two studied groups regarding post-delivery complain (P= 0.621, 0.102)

Table (6): Post delivery complain in the two studied groups.

| Post delivery complain | Group I | | Group II | | P value |
|------------------------|---------|------|----------|------|---------|
| | No | % | No | % | |
| No | 112 | 89.6 | 117 | 93.6 | 0.621 |
| Yes | 13 | 10.4 | 8 | 6.4 | 0.102 |
| Spotting | 8 | 61.5 | 4 | 50.0 | 0.071 |
| НМВ | 2 | 15.4 | 2 | 25.0 | 1.0 |
| Post coital bleeding | 3 | 23.1 | 2 | 25.0 | 0.92 |

Group I. cesarean section with bladder dissection

Group II: cesarean section without bladder dissection

 $\chi^2$  = Chi square-test



Figure (19): Post delivery complain in the two studied groups

# VII- Comparison between the two groups regarding incidence of postdelivery complaint and the type of contraceptive used

It was found that the highest incidence of complaint in both groups was found in cases with no contraceptive, followed by IUD user. There was statistical significant difference between two studied groups regarding complaint incidence in non contraceptive-user (P=0.036) (Table 7, Fig. 20)

Table (7): Relation between the incidence of post delivery complication and the type of contraceptive used.

| | Gro<br>"n= | up I<br>13" | Group II<br>"n=8" | | P value |
|-------------|------------|-------------|-------------------|------|---------|
| | No | % | No | % | |
| No | 7 | 46.2 | 5 | 62.5 | 0.036* |
| IUD | 3 | 23.1 | 2 | 25.0 | 0.521 |
| Pops | 1 | 7.7 | 0 | 0.0 | - |
| COCS | 1 | 7.7 | 0 | 0.0 | - |
| Depoprovera | 1 | 7.7 | 1 | 12.5 | 1.0 |



**Figure (20):** Relation between the incidence of post delivery complication and the type of contraceptive used.